CLINICAL TRIAL: NCT05661318
Title: Aswan Heart Centre - Ballana Heart Study
Brief Title: AHC Ballana Heart Study
Acronym: AHC-BHS
Status: Recruiting | Type: Observational
Sponsor: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AHC-BHS
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Genetic Predisposition to Disease
Keywords: genetics; Cardiovascular risks
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Risk Assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood for laboratory work up & whole genome sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BHS: Residents of Ballana from the 1,200 randomly selected households
  Interventions: Other: Risk assessment

INTERVENTIONS:
Other: Risk assessment — Collect clinical, laboratoary and genetics data from the participants after informed consent

SUMMARY:
This Study is designed to assess CVD incidence, prevalence, progression and related risk factors, including genetic background. It will provide an important base for all cardiovascular research activities in our centre and help in designing future studies and guide policy.

DETAILED DESCRIPTION:
Background Population-based longitudinal studies are a cornerstone in understanding current disease landscapes affecting communities and collecting reliable data to guide prevention and treatment strategies. In Egypt there is pressing need of collecting reliable data on cardiovascular disease (CVD) in defined populations.

Objectives Defining the cardiovascular phenotype, genotype as well as OMICS and risk factors for CVD in a defined population in Egypt with follow up for up to 30 years

Methods As a first step, a random representative sample of 1,200 households from the Ballana population will be created. Following inclusion, patients will be screened for their cardiovascular profile and followed up for changes in their profile and cardiovascular events continuously every year in high risk patients and every 3 years for the rest of the participants for a period of 30 years.

ELIGIBILITY:
Inclusion criteria:

* Residents of Ballana from the 1,200 randomly selected households
* Participants must have a valid National ID card
* Written informed consent

Exclusion criteria:

• Residents who are younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • Residents of Ballana from the 1,200 randomly selected households
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2055-01-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk assessment | 30 years

CONTACTS AND LOCATIONS:
Overall Officials: Magdi H Yacoub, FRS OM, Principal Investigator — Imperial College London, and Magdi Yacoub Heart Foundation
Locations (1):
- Aswan Heart Centre - Magdi Yacoub Heart Foundation, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keates AK, Mocumbi AO, Ntsekhe M, Sliwa K, Stewart S. Cardiovascular disease in Africa: epidemiological profile and challenges. Nat Rev Cardiol. 2017 May;14(5):273-293. doi: 10.1038/nrcardio.2017.19. Epub 2017 Feb 23. PMID 28230175